CLINICAL TRIAL: NCT00812214
Title: Treatment of Insomnia in Migraineurs With Eszopiclone (Lunesta™) and Its Effect on Sleep Time, Headache Frequency, and Daytime Functioning: a Randomized, Double-blind, Placebo-controlled, Parallel-group Pilot Study
Brief Title: Treatment of Insomnia in Migraineurs
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: MedVadis Research Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: ESRC024
Record Dates: First submitted 2008-12-18; First posted 2008-12-22 (Estimated); Results first posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-05

CONDITIONS: Insomnia; Migraine
Keywords: insomnia; migraine; eszopiclone; insomnia in migraineurs
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Migraine Disorders | interventions — Eszopiclone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Eszopiclone (Lunesta) 3mg (Experimental): Participants with IHS-II migraine with and/or without aura and with DSM-IV primary insomnia. They were treated for 6 weeks with 3mg eszopiclone, followed by a 2-week runout period. Participants came in for five visits: a screening visit, a randomization visit, a compliance visit, an end-treatment visit, and an exit/early termination visit.
  Interventions: Drug: eszopiclone
- Placebo (Placebo Comparator): Participants with IHS-II migraine with and/or without aura and with DSM-IV primary insomnia. They were treated for 6 weeks with placebo, followed by a 2-week runout period. Participants came in for five visits: a screening visit, a randomization visit, a compliance visit, an end-treatment visit, and an exit/early termination visit.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: eszopiclone — 3 mg tablet every night at bedtime
  Other Names: Lunesta
  Arms: Eszopiclone (Lunesta) 3mg
Drug: placebo — 1 tablet every night at bedtime
  Arms: Placebo

SUMMARY:
It is hypothesized that treating insomnia in migraineurs, many of whom also have tension headaches, prolongs total sleep time to the extent that it decreases overall headache frequency. Chronic headache sufferers also feel more tired during the day, undoubtedly affecting daytime functioning, which is hypothesized to improve as well with prolonged total sleep time.

DETAILED DESCRIPTION:
The objective of the study is to determine the effect of prolonging total sleep time in migraineurs with insomnia on overall headache frequency, daytime alertness, fatigue, and functioning. The prolongation of total sleep time is accomplished by bedtime administration of 3 mg eszopiclone (Lunesta™), compared with placebo through a parallel-group design.

ELIGIBILITY:
Inclusion criteria:

1. Men and women, 18 to 64 years of age (inclusive) with International Headache Society (IHS)-II migraine with/without aura and Diagnostic and Statistical Manual (DSM)-IV primary insomnia (sleep onset/sleep maintenance).
2. Migraine frequency is 4-12 times per month, with a maximum of 20 days with headache per month, for 1 month or longer prior to screening.
3. A usual, estimated total sleep time of 6½ hours per night or less, for 1 month or longer prior to screening, due to problems falling asleep, waking up during the night, or waking up early.

Exclusion criteria:

1. Abortive migraine treatment with schedule II-III opioids.
2. Use of caffeine-containing medications, prescription and non-prescription, not exceeding 10 days per month.
3. Preventive migraine treatment with tricyclics or anticonvulsants.
4. Treatment of insomnia with non-prescription medications, such as diphenhydramine, melatonin, or valerian, and prescription medications, such as hypnotics, barbiturates, benzodiazepines, sedating antihistamines, antidepressants, and antipsychotics.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2007-04; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Egilius LH Spierings, M.D., Ph.D., Principal Investigator — MedVadis Research Corporation

REFERENCES:
- [Result] Spierings EL, McAllister PJ, Bilchik TR. Efficacy of treatment of insomnia in migraineurs with eszopiclone (Lunesta(R)) and its effect on total sleep time, headache frequency, and daytime functioning: A randomized, double-blind, placebo-controlled, parallel-group, pilot study. Cranio. 2015 Apr;33(2):115-21. doi: 10.1179/0886963414Z.00000000084. Epub 2014 Oct 16. PMID 25323219

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 113 subjects were screened. 79 of them were randomized (69.9%). Of the 34 subjects who were not randomized, 8 were screen failures (23.5%), 17 were baseline failures (50.0%), 4 withdrew consent (11.8%), and 5 were lost to follow-up (14.7%).
Groups:
- Eszopiclone 3 mg: Participants with IHS-II migraine with and/or without aura and with DSM-IV primary insomnia. They were treated for 6 weeks with 3mg eszopiclone, followed by a 2-week runout period. Participants came in for five visits: a screening visit, a randomization visit, a compliance visit, an end-treatment visit, and an exit/early termination visit.
Period: Overall Study
Arm/Group | Eszopiclone 3 mg | Placebo
Started | 38 | 41
Completed | 35 | 40
Not Completed | 3 | 1
Not completed — Lost to Follow-up | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Eszopiclone 3 mg | Placebo | Total
Number analyzed (Participants) | 38 | 41 | 79
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 38 | 41 | 79
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.8 (11.1) | 45.0 (10.5) | 44.4 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 34 | 63
  Male | 9 | 7 | 16
Race/Ethnicity, Customized [Number; unit: percentage of participants] — Population: Baseline data only available for mITT participants (defined as all participants who took study medication at least 5 days per week for the first 2 weeks of the 6-week treatment period and provided the corresponding diary entries for sleep and headache)
  percentage of participants
    Caucasian: number analyzed (Participants) | 35 | 40 | 75
    Caucasian | 80 | 80 | 80
    Other: number analyzed (Participants) | 35 | 40 | 75
    Other | 20 | 20 | 20
Region of Enrollment [Number; unit: participants]
  United States | 38 | 41 | 79

OUTCOME MEASURES:

1. Primary Outcome: Total Sleep Time
Description: Participants were asked to record an estimated total time asleep on a daily basis. Nightly estimates were averaged over a 2 week period for baseline and 6 week period so that the total sleep time represents the average total time asleep each night.
Time Frame: Baseline, 6 weeks
Population: Modified ITT (defined as all participants who took study medication at least 5 days per week for the first 2 weeks of the 6-week treatment period and provided the corresponding diary entries for sleep and headache.)
Measure: Mean (Standard Deviation); unit: hours
Groups:
- Eszoplicone 3mg: Participants with IHS-II migraine with and/or without aura and with DSM-IV primary insomnia. They were treated for 6 weeks with 3mg eszopiclone, followed by a 2-week runout period. Participants came in for five visits: a screening visit, a randomization visit, a compliance visit, an end-treatment visit, and an exit/early termination visit.
Arm/Group | Eszoplicone 3mg | Placebo
Number analyzed (Participants) | 35 | 40
hours
  Baseline | 5.4 (0.8) | 5.5 (1.0)
  6 week average | 6.3 (0.9) | 6.1 (0.8)
Statistical Analysis 1: Comparison: Eszoplicone 3mg vs Placebo; The null hypothesis is that there is no difference in the 6 week average total sleep time; Test type: Superiority — For the purpose of the power calculation, it was assumed that the difference in total sleep time between the treatment groups is 40 minutes, with a standard deviation of 60. The pilot nature of the study allowed the use of alpha = 0.05 and beta = 0.2, with two-sided comparison, generating a required sample size of 37 subjects per arm; p = 0.33, t-test, 2 sided; two-tailed student's t-test for independent samples

2. Secondary Outcome: Nighttime Awakenings
Description: Participants were asked to keep a daily record. 6 week data were averaged over the 6 week period
Time Frame: Baseline, 6 weeks
Population: modified ITT
Measure: Mean (Standard Deviation); unit: awakenings/night
Groups:
- Eszopiclone 3mg: Participants with IHS-II migraine with and/or without aura and with DSM-IV primary insomnia. They were treated for 6 weeks with 3mg eszopiclone, followed by a 2-week runout period. Participants came in for five visits: a screening visit, a randomization visit, a compliance visit, an end-treatment visit, and an exit/early termination visit.
Arm/Group | Eszopiclone 3mg | Placebo
Number analyzed (Participants) | 35 | 40
awakenings/night
  Baseline | 2.4 (1.5) | 2.7 (1.3)
  6 weeks | 1.5 (1.1) | 2.2 (1.4)
Statistical Analysis 1: Comparison: Eszopiclone 3mg vs Placebo; The null hypothesis is that there is no difference between the eszopiclone and placebo groups in the number of awakenings/night at 6 weeks; Test type: Superiority; p = 0.03, t-test, 2 sided

3. Secondary Outcome: Nighttime Awakenings
Description: Participants were asked to keep a daily record.
  The average among weeks 1 and 2, weeks 3 and 4, and weeks 5 and 6 were taken, resulting in 3 averages, where the lowest average is reported as the minimum value of the full range, the middle average is reported as the median, and the highest average is reported as the maximum value of the full range
Time Frame: Measured every two weeks (1&2, 3&4, 5&6)
Population: modified ITT
Measure: Median (Full Range); unit: awakenings/night
Arm/Group | Eszopiclone 3mg | Placebo
Number analyzed (Participants) | 35 | 40
awakenings/night | 1.5 [1.5 to 1.6] | 2.1 [2.1 to 2.2]

4. Secondary Outcome: Quality of Sleep
Description: Participants were asked to keep a daily record. 6 week data were averaged over the 6 week period
  * Overall sleep quality was measured on a scale of 1=poor to 10=excellent.
  * Daytime alertness was measured on a scale of 1=not alert to 10=extremely alert.
  * Daytime fatigue was measured on a scale of 1=not tired to 10=extremely tired.
  * Daytime functioning was measured on a scale of 1=poor to 10=excellent.
Time Frame: Baseline, 6 weeks
Population: modified ITT
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Eszopiclone 3mg | Placebo
Number analyzed (Participants) | 35 | 40
score on a scale
  Overall sleep quality, Baseline | 5.1 (1.1) | 4.9 (1.1)
  Overall sleep quality, 6 weeks | 6.7 (1.2) | 6.2 (1.0)
  Daytime alertness, Baseline | 6.1 (1.1) | 6.0 (1.4)
  Daytime alertness, 6 weeks | 6.9 (1.3) | 6.6 (1.2)
  Daytime fatigue, Baseline | 5.2 (1.4) | 5.5 (1.5)
  Daytime fatigue, 6 weeks | 4.3 (1.4) | 5.0 (1.5)
  Daytime functioning, Baseline | 6.5 (1.2) | 6.3 (1.5)
  Daytime functioning, 6 weeks | 7.0 (1.3) | 6.9 (1.3)
Statistical Analysis 1: Comparison: Eszopiclone 3mg vs Placebo; Null hypothesis is that there is no difference between Eszopiclone and placebo groups in sleep quality averaged over 6 weeks of treatment; Test type: Superiority; p = 0.1, t-test, 2 sided
Statistical Analysis 2: Comparison: Eszopiclone 3mg vs Placebo; Null hypothesis is that there is no difference between Eszopiclone and placebo groups in daytime alertness averaged over 6 weeks of treatment; Test type: Superiority; p = 0.29, t-test, 2 sided
Statistical Analysis 3: Comparison: Eszopiclone 3mg vs Placebo; Null hypothesis is that there is no difference between Eszopiclone and placebo groups in daytime fatigue averaged over 6 weeks of treatment; Test type: Superiority; p = 0.05, t-test, 2 sided
Statistical Analysis 4: Comparison: Eszopiclone 3mg vs Placebo; Null hypothesis is that there is no difference between Eszopiclone and placebo groups in daytime functioning averaged over 6 weeks of treatment; Test type: Superiority; p = 0.76, t-test, 2 sided

5. Secondary Outcome: Daytime Fatigue
Description: Participants were asked to keep a daily record.
  * Daytime fatigue was measured on a scale of 1=not tired to 10=extremely tired.
  The average among weeks 1 and 2, weeks 3 and 4, and weeks 5 and 6 were taken, resulting in 3 averages, where the lowest average is reported as the minimum value of the full range, the middle average is reported as the median, and the highest average is reported as the maximum value of the full range
Time Frame: Measured every two weeks (1&2, 3&4, 5&6)
Population: modified ITT
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Eszopiclone 3mg | Placebo
Number analyzed (Participants) | 35 | 40
score on a scale | 4.3 [4.2 to 4.4] | 4.8 [4.8 to 5.2]

6. Secondary Outcome: Headache Frequency
Description: Number of days per week in which a participant had a headache. Participants were asked to keep a daily record. 6 week data were averaged over the 6 week period
Time Frame: Baseline, 6 weeks
Population: modified ITT
Measure: Mean (Standard Deviation); unit: days/week
Arm/Group | Eszopiclone 3mg | Placebo
Number analyzed (Participants) | 35 | 40
days/week
  Baseline | 2.9 (1.2) | 3.1 (1.2)
  6 weeks | 2.5 (1.3) | 2.5 (1.4)
Statistical Analysis 1: Comparison: Eszopiclone 3mg vs Placebo; The null hypothesis is that there is no difference in average days/week between eszopiclone and placebo groups at 6 weeks; Test type: Superiority; p = 0.89, t-test, 2 sided

7. Secondary Outcome: Headache Duration
Description: Participants were asked to keep a daily record. 6 week data were averaged over the 6 week period
Time Frame: Baseline, 6 weeks
Population: modified ITT
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Eszopiclone 3mg | Placebo
Number analyzed (Participants) | 35 | 40
hours
  Baseline | 4.0 (2.3) | 3.7 (2.2)
  6 weeks | 3.9 (1.8) | 3.8 (2.2)
Statistical Analysis 1: Comparison: Eszopiclone 3mg vs Placebo; The null hypothesis is that there is no difference in headache duration between eszopiclone and placebo groups at 6 weeks; Test type: Superiority; p = 0.98, t-test, 2 sided

8. Secondary Outcome: Headache Intensity
Description: Participants were asked to keep a daily record. 6 week data were averaged over the 6 week period
  * Headache intensity was measured on a scale of 1=not intense to 10=worst headache possible
Time Frame: Baseline, 6 weeks
Population: modified ITT
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Eszopiclone 3mg | Placebo
Number analyzed (Participants) | 35 | 40
score on a scale
  Baseline | 5.6 (2.3) | 5.3 (1.6)
  6 weeks | 5.5 (2.0) | 5.6 (1.8)
Statistical Analysis 1: Comparison: Eszopiclone 3mg vs Placebo; The null hypothesis is that there is no difference in headache intensity between eszopiclone and placebo groups at 6 weeks; Test type: Superiority; p = 0.82, t-test, 2 sided

ADVERSE EVENTS:
Description: All participants who were randomized
Arm/Group | Eszopiclone 3mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/41
Other Adverse Events (participants affected / at risk) | 0/38 | 0/41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes